CLINICAL TRIAL: NCT01866020
Title: Diagnosis of Invasive Pulmonary Aspergillosis (IPA) in Critically Ill Patients - a Prospective Clinical Trial in the Department of Intensive Care, University Medical Center Hamburg-Eppendorf (UKE)
Brief Title: Diagnosis of Invasive Pulmonary Aspergillosis (IPA) in Critically Ill Patients
Acronym: DipA
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: DipA
Record Dates: First submitted 2013-05-27; First posted 2013-05-31 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Survival After IPA; Risk Factors for IPA
Keywords: aspergillosis; fungal infection; ICU
MeSH Terms: conditions — Aspergillosis; Mycoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Invasive pulmonary aspergillosis (IPA) is difficult to diagnose and remains a cause of high morbidity and mortality in critically ill patients in the ICU. Accepted diagnostic protocols for haemato-oncological patients are not applicable for critically ill patients in ICUs. Definitive discrimination between aspergillic colonisation and IPA often depends on the clinical experience of the treating physician, evaluating clinical signs, co-morbidities, and course of the disease. Life saving treatment with the first line antimycotic Voriconazol (Vfend®) can only be initiated after diagnosis of IPA.

In this prospective clinical trial the investigators aim to structure, optimize and fast track the diagnostic pathway of IPA in critically ill patients treated in our ICU-department.

DETAILED DESCRIPTION:
Invasive pulmonary aspergillosis (IPA) is difficult to diagnose and remains a cause of high morbidity and mortality in critically ill patients in the ICU. The number of patients with positive Aspergillus culture or galactomannan test in respiratory fluids is increasing every year. In 2007 our Department tested 21 patients positive for Aspergillus, in 2009 it were 49 and last year (2011) the investigators found 59 patients to be positive in our 10 multidisciplinary ICUs. Accepted diagnostic protocols for haemato-oncological patients are not applicable for critically ill patients in ICUs. Halo signs, a typical radiological indication for IPA, can be found in haematological patients, but in patients in the ICU these signs are likely to be masked by pneumonic infiltrations due to ventilator induced lung injury and pneumonia. Microbiological diagnostics, like quantification of galactomannan in bronchoalveolar lavage specimens, change upon antibiotic treatment. It can be false positive in patients treated with beta-lactam antibiotics. Definitive discrimination between aspergillic colonisation and IPA often depends on the clinical experience of the treating physician, evaluating clinical signs, co-morbidities, and course of the disease. Life saving treatment with the first line antimycotic Voriconazol (Vfend®) can only be initiated after diagnosis of IPA.

In this prospective clinical trial the investigators aim to structure, optimize and fast track the diagnostic pathway of IPA in critically ill patients treated in our ICU-department. After successful diagnosis, primary endpoints of this study will be 28-day mortality and duration of the ICU stay. Secondary endpoints will include differences in antimycotic treatments, ventilation time and type of ventilation, co - morbidities and treatment costs between patients in the colonisation and IPA group.

Adult patients treated in one of our ten multidisciplinary ICUs with either positive respiratory fluid cultures for Aspergillus species or positive galactomannan test will be prospectively enrolled. During the 18 month enrollment period (January 2013 until July 2014) the investigators plan to screen all critically ill patients and enroll a minimum of 60 patients, which represents the expected number of patients diagnosed with an IPA in the proposed time frame. In agreement with our standard operating procedure, all study patients will be routinely subjected to the following examinations, tests and receive diagnostic interventions, but the investigator does not assign specific interventions to the patients of the study. A bronchoalveolar lavage, will be performed by a senior pulmonologist, to identify typical Aspergillus plaques and to obtain sufficient material for microbiological analysis (galactomannan test + polymerase chain reaction (PCR)). Blood samples for a galactomannan test will be drawn additionally. The galactomannan tests will be repeated weekly as long as the infection symptoms persist. Furthermore, patients will be subjected to high-resolution computer tomography of the thorax. Clinical and diagnostic data from all patients will be collected in a centralized database for subsequent analysis in this study.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* positive aspergillus culture in respiratory tract sample OR
* positive aspergillus galactomannan in respiratory tract sample

Exclusion Criteria:

* no inform consent
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
death after 6 month | 6 month
  we follow the patients after 6 month

SECONDARY OUTCOMES:
death after 28 days | 28 days
  we follow the patients for 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Maria Metschke, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

REFERENCES:
- [Derived] Schroeder M, Simon M, Katchanov J, Wijaya C, Rohde H, Christner M, Laqmani A, Wichmann D, Fuhrmann V, Kluge S. Does galactomannan testing increase diagnostic accuracy for IPA in the ICU? A prospective observational study. Crit Care. 2016 May 10;20(1):139. doi: 10.1186/s13054-016-1326-1. PMID 27160692